CLINICAL TRIAL: NCT04623151
Title: Manipulating Narrative Presentations of Information to Encourage Good Foot Care Practice in People With and Without Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chichester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UOCMRPHDS3
Record Dates: First submitted 2017-10-16; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot; Health Behavior; Foot Diseases
Keywords: Foot care; narrative; diabetes; health behaviour; health psychology
MeSH Terms: conditions — Diabetic Foot; Health Behavior; Foot Diseases; Narration; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 1. Online leaflet about foot care in a narrative format
  2. Online leaflet about foot care in a non-narrative format
  3. No leaflet (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online leaflet in narrative format (Experimental)
  Interventions: Behavioral: Online leaflet about foot care
- Online leaflet in non-narrative format (Active Comparator)
  Interventions: Behavioral: Online leaflet about foot care
- No leaflet (control) (No Intervention)

INTERVENTIONS:
Behavioral: Online leaflet about foot care — Short text-based leaflet about foot care, presented online
  Arms: Online leaflet in narrative format; Online leaflet in non-narrative format

SUMMARY:
The study explores the role of health messages (narrative, non-narrative vs. control condition [no message]) to enhance good foot care practices among people with diabetes and the general population.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age at the time of consent;
* able to read and speak the English language;
* able and willing to give written informed consent prior to study entry;
* able to complete the protocol requirements

Exclusion Criteria:

* has a cognitive impairment or acute psychopathology (self-reported formal diagnoses of down syndrome, traumatic brain injury, brain tumour, autism, dementia, schizophrenia, and/or schizoaffective disorder), ie that which could interfere with his or her ability to provide written consent and complete the study
* has taken part in any other research on foot care with the University of Chichester in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
5-item Foot Care Detection Behaviour Scale | 1 week
  Questionnaire asking participants how many days in the past 7 they have checked their feet to detect cuts, blisters, sores, calluses, and red patches

CONTACTS AND LOCATIONS:
Overall Officials: Susan Churchill, PhD, Study Director — University of Chichester
Locations (1):
- University of Chichester, Chichester, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the study team

REFERENCES:
- See also: Online survey — https://chichpscyh.eu.qualtrics.com/jfe/form/SV_eCF14PjJGVN0nGt